CLINICAL TRIAL: NCT01485367
Title: Phase II Pilot Study to Evaluate The Efficacy of Adapalene 0.3% for Use in The Prevention and Treatment of Senile Purpura
Brief Title: A Pilot Study to Evaluate The Efficacy of Adapalene 0.3% for Use in the Prevention and Treatment of Senile Purpura
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Multispecialty Aesthetic Clinical Research Organization (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AD3001
Record Dates: First submitted 2011-11-17; First posted 2011-12-05 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Senile Purpura
Keywords: Senile Purpura; Adapalene 0.3%

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapalene gel 0.3% (Active Comparator): All odd numbered subjects will receive treatment to the left arm. The untreated arm will serve as an intrapatient control and will be evaluated separately from the treated arm for signs of purpura.
  Interventions: Drug: adapalene gel 0.3%
- Adapalene gel 0.3 % (Active Comparator): All even numbered subjects will receive treatment to the right arm. The untreated arm will serve as an intrapatient control and will be evaluated separately from the treated arm for signs of purpura.
  Interventions: Drug: adapalene gel 0.3%

INTERVENTIONS:
Drug: adapalene gel 0.3% — A pea size drop of Adapalene gel 0.3% will be applied to the odd numbered subjects on the left dorsal hand & extensor forearm. A pea size drop of Adapalene gel 0.3% will be applied to the even numbered subjects on the right dorsal hand & extensor forearm. The randomized area will be cleansed with Cetaphil Gentle Cleanser before applying the study medication. All subjects will apply sunscreen with zinc oxide in the morning to both the right & left forearms.
  Other Names: Differin gel 0.3%

SUMMARY:
This is an open label 6 month pilot study for male and female participants over the age of 52 that desire treatment and prevention of senile purpura of the forearms.

This study will be evaluating the effects of Adapalene 0.3% for the use in the treatment and prevention of senile purpura.

DETAILED DESCRIPTION:
This is a new potential use for the product Adapalene 0.3%, which is currently an FDA approved topical treatment used for the treatment of acne.

Senile purpura is a common sign of aging that appears in the form of dark blotches on the skin and is caused by bruising.

Older adults tend to be more prone to bruising, since as people age, their skin becomes thinner and more fragile.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 52 years of age with signs of senile purpura on either the right or left (or both) dorsal hand & extensor forearm and desire treatment for this condition that is associated with aging.
* Women who have had hysterectomies, tubal ligations or who are post-menopausal for at least one year prior to the study may be enrolled. Women of childbearing potential who are not pregnant, not planning to become pregnant during the study period, and not lactating may be enrolled if they are using a medically accepted contraceptive program initiated at least one month prior to study entry and continued during the study.
* Subject is willing to comply with study instructions and return to the clinic for required visits.
* Subject is able to understand and has signed an IRB approved informed consent form including consent for photography.

Exclusion Criteria:

* All subjects on coumadin, heparin, plavix, supplemental herbs, vitamin E, empirin, fiorinal, norgesic, forte, percodan, robaxin, nuprin, ansaid, anaprox, clinoril, dolobid, feldene, naprosyn, voltaren, fish oil, oral steroids, or daily use of aspirin, Motrin, or Advil. (PRN usage not excluded)
* Prior treatment with any systemic immunosuppressive therapy including but not limited to chemotherapy agents or corticosteroids within 3 months of study enrollment is prohibited.
* Clotting abnormalities as determined by screening labs
* Any history of a stroke or unstable heart disease
* Participation in another clinical trial with exposure to any investigational agent within 30 days prior to Screening Visit.
* Any condition the Investigator believes would interfere with subject's ability to provide informed consent, comply with study instruction, or which might confound the interpretation of the study results or put the subject at undue risk.
* Subject is pregnant, breastfeeding or planning a pregnancy during the study.
* Subject is unable to communicate or cooperate with the Investigator due to a language barrier (non-English speaking).
* Subjects who are allergic to adapalene or the ingredients in the gel.

Min Age: 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Show the clinical benefit of daily application of Adapalene 0.3% in decreasing the signs of senile purpura | Up to 6 months
  To evaluate and document the degree of aesthetic results of subjects with senile purpura using the MACRO MD Purpura Lesion Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hamilton, MD, Principal Investigator — Multispecialty Aesthetic Clinical Research Organization
Locations (1):
- Multispecialty Aesthetic Clinical Research Organization, Woodland Hills, California, United States